CLINICAL TRIAL: NCT06574672
Title: Impact of an Embedded Palliative Care and Hospice Practitioner in the Medical ICU
Brief Title: Embedded Palliative Care in the MICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Stephen Wen-Yan Chi, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 202406143
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness; End of Life; Quality of Life
Keywords: Palliative Care; Hospice; Medical ICU
MeSH Terms: conditions — Critical Illness; Death | interventions — Health Records, Personal

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prospective Hospice and Palliative Care Intervention (Experimental): This arm comprises patients admitted to the specific medical intensive care unit in which the hospice and palliative care practitioner is currently active. This will include all patients admitted to a single medical intensive care unit during the anticipated first half of the intervention timeframe, followed by all patients admitted to both medical intensive care units during the second half of the intervention timeframe.
  Interventions: Other: Embedded Hospice and Palliative Care Practitioner
- Prospective Standard of Care (Active Comparator): This arm comprises patients admitted to the medical intensive care unit in which the hospice and palliative care practitioner is not currently active, but which may experience a group effect due to the study's ongoing enrollment and the practitioner's presence. This will include all patients admitted to a single medical intensive care unit during the anticipated first half of the intervention timeframe, prior to the practitioner becoming active in both intensive care units.
  Interventions: Other: Embedded Hospice and Palliative Care Practitioner (Group Effect)
- Historical Controls (Placebo Comparator): This arm comprises historical patients admitted to the medical intensive care units in the year prior to study enrollment.
  Interventions: Other: None (Historical)

INTERVENTIONS:
Other: Embedded Hospice and Palliative Care Practitioner — The hospice and palliative care practitioner will be embedded in one medical intensive care unit for the first half of the study timeframe, after which the practitioner will expand to both medical intensive care units. While active in a medical intensive care unit, the practitioner will proactively trigger palliative care consultations based on clinical criteria and estimated mortality risk, in addition to providing immediate availability for standard-of-care hospice or palliative care consultations.
  Arms: Prospective Hospice and Palliative Care Intervention
Other: Embedded Hospice and Palliative Care Practitioner (Group Effect) — While the hospice and palliative care practitioner is active in one medical intensive care unit with respect to triggering consultations, the other medical intensive care unit can still utilize the practitioner's services for standard-of-care hospice or palliative care consultations.
  Arms: Prospective Standard of Care
Other: None (Historical) — This control arm includes historical patients admitted to the medical intensive care units prior to the study's enrollment timeframe.
  Arms: Historical Controls

SUMMARY:
The goal of this study is to investigate whether embedding a hospice and palliative care practitioner within a medical intensive care unit will improve patient outcomes and healthcare usage. The practitioner will work solely within the medical intensive care units and offer timely as well as proactive consultations based on clinical criteria and estimated mortality risk. The study team will compare patients seen by the practitioner to patients in an adjacent ICU and historical patients to determine whether patient care is improved by this intervention.

DETAILED DESCRIPTION:
The study goal is to determine whether an embedded palliative care practitioner in the medical ICU improves patient outcomes, palliative care/hospice utilization, and healthcare quality metrics. The medical ICUs included in this study are comprised of two geographically co-located units that provide care for medically complex patients from a large tertiary referral area. Palliative care services are currently available as a consultative service at the ICU clinicians' discretion for patients with palliative needs such as complex goals of care, advanced symptom management, or chronic critical illness. Under the current consultation model, palliative care consultation is requested in a minority of critically ill patients and consults occur on average 5-14 days after a patient's admission. Hospice services are similarly available on a consultative basis for patients that the primary team has determined are suitable for hospice, however, logistical limitations of hospice consultation may lead to delays in inpatient hospice transfers and home hospice discharges.

This study's intervention is to embed a palliative care/hospice practitioner within the medical ICUs as a dedicated palliative care and hospice consultant who will offer proactively triggered palliative care consultations early in a patient's ICU stay as well as immediate availability for standard-of-care palliative care and hospice consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical intensive care units at a tertiary referral center
* Patients must be at least 18 years of age

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
ICU Length of Stay | From date of enrollment until hospital discharge, assessed up to 1 year
  Length of stay in any intensive care unit during the hospitalization
Code Status De-escalation | From date of enrollment until hospital discharge, assessed up to 1 year
  Frequency of changes in code status to limited code or comfort measures only

SECONDARY OUTCOMES:
Presence of Advance Care Planning Documentation during Current Admission | From date of enrollment until hospital discharge, assessed up to 1 year
  Documentation of advance directives, limitations in life-sustaining treatments, or code status that is newly created during the active hospital admission
Hospice Consultation | From date of enrollment until hospital discharge, assessed up to 1 year
  Frequency of Hospice consultations
Hospice Enrollment | From date of enrollment until hospital discharge, assessed up to 1 year
  Frequency of discharge or transition to hospice during or immediately following the hospital stay
Palliative Care Consultation | From date of enrollment until hospital discharge, assessed up to 1 year
  Frequency of Palliative Care consultations
Time to change in code status, advance care planning documentation, palliative care consultation, and hospice consultation | From date of enrollment until hospital discharge, assessed up to 1 year
  Time in days to the first occurrence of the above outcomes
Inpatient Hospice Duration | From date of enrollment until hospital or hospice discharge, assessed up to 1 year
  Days while patients are enrolled in inpatient hospice (GIP)
Location of discharge disposition | From date of enrollment until hospital discharge, assessed up to 1 year
  Discharge disposition to home, skilled nursing facility, long term acute care facility, inpatient rehabilitation, etc.
Hospital Length of Stay | From date of enrollment until hospital discharge, assessed up to 1 year
  Length of hospital stay in days
Mortality Index (Vizient) | From date of enrollment until hospital discharge, assessed up to 1 year
  Mortality index as calculated by Vizient
Length of Stay Index (Vizient) | From date of enrollment until hospital discharge, assessed up to 1 year
  Length of stay index as calculated by Vizient
Operating cost in dollars, including departmental breakdown | Assessed six months following discharge
  Hospital operating cost for each patient, including departmental breakdown such as ICU, pharmacy, procedural, operating room, etc.
Mechanical Ventilation Duration | From date of enrollment until hospital discharge, assessed up to 1 year
  Days on mechanical ventilation
Vasopressor Utilization | From date of enrollment until hospital discharge, assessed up to 1 year
  Days on vasopressors
Hospital Mortality | From date of enrollment until hospital discharge, assessed up to 1 year
  Inpatient all-cause mortality
30-Day Mortality | Assessed 30 days after hospital admission
  All-cause mortality within 30 days of hospital admission
30-day Emergency Room Visit | Assessed 30 days after hospital discharge
  Emergency Room encounter in the same healthcare system within 30 days of discharge
30-day Readmission | Assessed 30 days after hospital discharge
  Hospital readmission in the same healthcare system within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chi, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslakson R, Cheng J, Vollenweider D, Galusca D, Smith TJ, Pronovost PJ. Evidence-based palliative care in the intensive care unit: a systematic review of interventions. J Palliat Med. 2014 Feb;17(2):219-35. doi: 10.1089/jpm.2013.0409. PMID 24517300
- [Background] Khandelwal N, Kross EK, Engelberg RA, Coe NB, Long AC, Curtis JR. Estimating the effect of palliative care interventions and advance care planning on ICU utilization: a systematic review. Crit Care Med. 2015 May;43(5):1102-11. doi: 10.1097/CCM.0000000000000852. PMID 25574794
- [Background] Kyeremanteng K, Gagnon LP, Thavorn K, Heyland D, D'Egidio G. The Impact of Palliative Care Consultation in the ICU on Length of Stay: A Systematic Review and Cost Evaluation. J Intensive Care Med. 2018 Jun;33(6):346-353. doi: 10.1177/0885066616664329. Epub 2016 Aug 31. PMID 27582396
- [Background] Braus N, Campbell TC, Kwekkeboom KL, Ferguson S, Harvey C, Krupp AE, Lohmeier T, Repplinger MD, Westergaard RP, Jacobs EA, Roberts KF, Ehlenbach WJ. Prospective study of a proactive palliative care rounding intervention in a medical ICU. Intensive Care Med. 2016 Jan;42(1):54-62. doi: 10.1007/s00134-015-4098-1. Epub 2015 Nov 10. PMID 26556622
- [Background] Helgeson SA, Burnside RC, Robinson MT, Mack RC, Ball CT, Guru PK, Moss JE. Early Versus Usual Palliative Care Consultation in the Intensive Care Unit. Am J Hosp Palliat Care. 2023 May;40(5):544-551. doi: 10.1177/10499091221115732. Epub 2022 Jul 14. PMID 35833450
- [Background] Ma J, Chi S, Buettner B, Pollard K, Muir M, Kolekar C, Al-Hammadi N, Chen L, Kollef M, Dans M. Early Palliative Care Consultation in the Medical ICU: A Cluster Randomized Crossover Trial. Crit Care Med. 2019 Dec;47(12):1707-1715. doi: 10.1097/CCM.0000000000004016. PMID 31609772
- [Background] Chi S, Kim S, Reuter M, Ponzillo K, Oliver DP, Foraker R, Heard K, Liu J, Pitzer K, White P, Moore N. Advanced Care Planning for Hospitalized Patients Following Clinician Notification of Patient Mortality by a Machine Learning Algorithm. JAMA Netw Open. 2023 Apr 3;6(4):e238795. doi: 10.1001/jamanetworkopen.2023.8795. PMID 37071421

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT06574672/SAP_000.pdf